CLINICAL TRIAL: NCT01666535
Title: Effect of Influenza Vaccination Timing on Immune Response in Patients With Inflammatory Bowel Disease on Infliximab Therapy: A Randomized Equivalence Trial
Brief Title: Infliximab IBD Influenza Vaccine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer deBruyn, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REMICADEIBD4010
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: Influenza vaccine; Immune response; Remicade (infliximab); Inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccination Timing #1 (Other): Influenza vaccination administered on the same day as infliximab administration (Day 0 to 4).
  Interventions: Biological: Influenza vaccination
- Influenza vaccination Timing #2 (Other): Influenza vaccination administered at the mid-point between infliximab infusions (Day 21 to 28)
  Interventions: Biological: Influenza vaccination

INTERVENTIONS:
Biological: Influenza vaccination

SUMMARY:
The investigators will compare the immunogenicity of influenza vaccine in adults and children with inflammatory bowel disease by timing of vaccine in relation to maintenance infliximab dosing. The primary objective is to compare the proportion of IBD patients on maintenance infliximab who mount serologic protection to each component of the influenza vaccination between patients vaccinated on day of infliximab infusion (Day 0 to 4) and patients vaccinated at the mid-point between infliximab infusions (Day 21 to 28). Serologic protection will be defined by a hemagglutination-inhibition titer ≥ 1:40. The secondary objective is to compare the proportion of IBD patients who mount an immunogenic response (≥ 4-fold increase from pre to post-vaccination titer) to each component of the influenza vaccination between patients vaccinated on day of infliximab infusion and those vaccinated at the mid-point.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD established by accepted criteria
* On maintenance infliximab administered every 6 to 8 weeks (already received at least 6 weeks of infliximab)
* Between ages 9 and 60 years

Exclusion Criteria:

1. Pregnancy
2. Hypersensitivity reaction to previous dose of influenza vaccine
3. Known hypersensitivity to eggs or chicken or other components of influenza vaccine

Ages: 9 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Serologic protection | 28 days ± 3 days after influenza vaccination
  To compare the proportion of IBD patients on maintenance infliximab who mount serologic protection to each component of the influenza vaccination between patients vaccinated on day of infliximab infusion (Day 0 to 4) and patients vaccinated at the mid-point between infliximab infusions (Day 21 to 28). Serologic protection will be defined by a hemagglutination-inhibition titer ≥ 1:40.

SECONDARY OUTCOMES:
Immunogenic response | 28 days ± 3 days after influenza vaccination
  To compare the proportion of IBD patients on maintenance infliximab who mount an immunogenic response to each component of the influenza vaccination between patients vaccinated on day of infliximab infusion (Day 0 to 4) and patients vaccinated at the mid-point between infliximab infusions (Day 21 to 28). Immunogenicity will be defined as a fourfold or greater differences in titer between pre and post-vaccination sera.

OTHER OUTCOMES:
Number of participants with serious adverse events | 3 days post vaccination
  To evaluate the number of participants with early serious adverse reactions (≤ 3 days post-vaccination)
Change in disease activity from baseline | Four week post-vaccination
  To evaluate the change in disease activity score from baseline using the validated instruments of the Pediatric Ulcerative Colitis Activity Index for participants with Ulcerative Coltiis and the Harvey Bradshaw Index for participants with Crohn's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer deBruyn, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada